CLINICAL TRIAL: NCT04059302
Title: Internet Cognitive Behavioral Therapy for Insomnia to Prevent Cardiovascular Disease
Acronym: STOPCVD
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Intervention services were suspended and then unavailable.
Sponsor: Megan Petrov (Other)
Responsible Party: Sponsor-Investigator, Megan Petrov, Assistant Professor, Arizona State University
Organization: Arizona State University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY00004470
Record Dates: First submitted 2019-07-10; First posted 2019-08-16 (Actual); Last update posted 2023-07-19 (Actual); Status verified 2023-07

CONDITIONS: Insomnia Chronic; Subclinical Disease and/or Syndrome
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The ultra sound technician that will be evaluating the primary outcome measures will be blinded to participant condition.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Online CBT-I (Experimental): Fully-automated, internet-delivered cognitive behavioral therapy for insomnia program that consists of 6 therapy cores delivered weekly over 6 weeks.
  Interventions: Behavioral: Internet-delivered Cognitive Behavioral Therapy for Insomnia
- Wait-List Control (No Intervention): Wait-list control group will receive no intervention until after the trial period is completed. During the trial period they will complete all study assessments, but receive no active treatment.

INTERVENTIONS:
Behavioral: Internet-delivered Cognitive Behavioral Therapy for Insomnia — The therapy consists of 6 modules or 'cores' that are introduced on a weekly basis. The cores are designed to decrease sleep-inhibiting cognitions and behaviors, and to alter sleep-wake schedules.
  Arms: Online CBT-I

SUMMARY:
This randomized controlled trial will test the efficacy of online cognitive-behavioral therapy for insomnia (CBT-I) to improve markers of subclinical cardiovascular disease risk among middle aged adults (40-64 years) with chronic insomnia who are at moderate-to-high risk for cardiovascular disease. Multiple trials have revealed face to face and digital CBT-I improves insomnia symptoms and associated daytime functioning. However, CBT-I has not been tested as a primary prevention intervention to reduce risk for CVD. Mid-life adults are a high-risk group for the emergence of CVD with detrimental consequences pervading into older adulthood including reduced quality of life and greater health care costs. The investigators will evaluate whether online CBT-I affects vascular and cardiac function and structure at post-treatment and 8-week follow-up in a community-based sample.

Hypothesis 1: Online CBT-I will improve indices of cardiovascular function and structure compared to a wait-list control group at post-treatment.

Hypothesis 2: Improvements in indices of cardiovascular function and structure will be maintained at 8-week follow-up in the online CBT-I group.

DETAILED DESCRIPTION:
In this randomized controlled trial, comparing internet-delivered cognitive behavioral therapy for insomnia (CBT-I) to a wait-list control group on pre-post trial changes in indices of cardiovascular structure and function among community-based middle-aged adults with insomnia and moderate-to-high risk for cardiovascular disease, the investigators will recruit and enroll 38 participants.

Initial screening will be conducted with an online survey. If they meet preliminary study criteria, then research staff will contact the participant to schedule an in-person, baseline assessment visit. They will be instructed that they must meet fasting requirements prior to this visit to obtain accurate cardiovascular physiology measurement.

At the baseline assessment visit, the participants will undergo the informed consent process, complete questionnaire inquiring about medical, mental, and sleep health history, undergo a brief physical (vital signs, height, weight), and complete cardiovascular physiology assessment. If the participants remain eligible after these assessment, then the pariticpants will receive orientation on how to complete an online sleep diary while simultaneously wearing a wrist actigraph to track sleep and activity for the next 7 nights. This procedure is for baseline assessment. It will not be used to further screen participants.

Once the participants complete this baseline sleep assessment, then they will randomly assigned to either immediate treatment with internet delivered CBT-I or a wait-list control group. The intervention group will receive an email with their own personal subscription to the online CBT-I program. Both groups will continue to wear the wrist actigraph for the duration of the trial. The immediate CBT-I group will complete sleep diaries within the online therapy program throughout the trial, whereas the wait-list control group will complete email-delivered, online sleep diaries from study staff throughout the trial.

The online Cognitive Behavioral Therapy for Insomnia intervention is based in a standardized, manualized treatment designed to decrease sleep-inhibiting cognitions and behaviors, and to alter sleep-wake schedules. This fully automated therapy tailors its program features according to sleep diary data inputs. The therapy will consist of CBTI-I components: stimulus control therapy, sleep restriction therapy, cognitive therapy, and sleep education. The first week of treatment will solely focus on sleep education and completion of sleep logs.

Upon completion of the treatment period, all participants will complete one more week of sleep diaries and wearing the wrist actigraph. The participants also will be scheduled to attend their post-treatment/trial in-person visit for assessment and to return the actigraph. Participants will complete questionnaires and undergo cardiovascular physiological assessment.

After this post-treatment visit, the wait-list control group will receive their subscription of the internet-delivered CBT-I program.

Participants randomly assigned to immediate internet delivered CBT-I will be scheduled for an 8-week follow-up visit during which they will once again complete outcome questionnaires and cardiovascular physiological assessment.

ELIGIBILITY:
Inclusion Criteria:

* All participants must be 40-64 years of age, able to understand English, score 10 or higher on the Insomnia Severity Index, >30 minutes nocturnal wakefulness (sleep onset latency or wake after sleep onset) for at least 3 nights per week, meet International Classification of Sleep Disorders-III [ISCD-3] diagnostic criteria for an insomnia disorder (see below), have a family history of cardiovascular disease, and screen positive for impaired FMD (< 7% difference between brachial artery diameter before and after occlusion).

ICSD-3 criteria for insomnia disorder:

A. The patient reports one or more of the following:

1. Difficulty initiating sleep.
2. Difficulty maintaining sleep.
3. Waking up earlier than desired.

B. The patient reports, one or more of the following related to the nighttime sleep difficulty:

1. Fatigue/malaise.
2. Attention, concentration, or memory impairment.
3. Impaired social, family, occupational, or academic performance.
4. Mood disturbance/irritability.
5. Daytime sleepiness.
6. Behavioral problems (e.g., hyperactivity, impulsivity, aggression).
7. Reduced motivation/energy/initiative.
8. Proneness for errors/accidents.
9. Concerns about or dissatisfaction with sleep. C. The reported sleep/wake complaints cannot be explained purely by inadequate opportunity (i.e., enough time is allotted for sleep) or inadequate circumstances (i.e., the environment is safe, dark, quiet, and comfortable) for sleep.

D. The sleep disturbance and associated daytime symptoms occur at least three times per week.

E. The sleep disturbance and associated daytime symptoms have been present for at least three months F. The sleep/wake difficulty is not better explained by another sleep disorder.

Exclusion Criteria:

* Participant will be excluded if they screen positive using retrospective questionnaires for other sleep disorders (see appendix of questionnaires), are involved in shift work, have a personal history of cardiovascular disease (i.e., myocardial infarction, atrial fibrillation, stroke, transient ischemic attack, diabetes, peripheral vascular disease), untreated Stage 2 hypertension (i.e., systolic blood pressure ≥ 160; diastolic blood pressure ≥ 100), current or diagnosis of psychiatric disorder within the past six months (including psychotic, mood, and anxiety disorders), start of psychotherapy within the past 6 months, clinically significant depressive symptoms as measured by a score of 10 or greater on the Center for Epidemiologic Studies Depression (CESD)-10 Revised scale, current or previous history of behavioral interventions for insomnia, currently smoking or using other nicotine products, excessive use of caffeine (>4 cups/day) or alcohol (>2 drinks/day), current and frequent use (2+ per week) of sleep medications, and engaging in vigorous exercise 75+ minutes/week. Women who are peri-menopausal, pregnant, breastfeeding, or trying to become pregnant will also be excluded.

Ages: 40 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2019-09-20 (Actual); Primary Completion 2021-07-15 (Actual); Study Completion 2021-07-15 (Actual)

PRIMARY OUTCOMES:
Change in Baseline to Post-Treatment endothelial-dependent dilation of the brachial artery (FMD) | Baseline; Post-treatment: 7 weeks after treatment initiation
  A non-invasive assessment of the ability of the brachial (upper arm) artery to dilate in response to an increase in blood flow, and is assessed using ultrasound.

SECONDARY OUTCOMES:
Change in baseline to post-treatment carotid-femoral pulse wave velocity (a measure of aortic stiffness) | Baseline; Post-treatment: 7 weeks after treatment initiation
  Pulse wave velocity = distance/time in m/s. Distance is 80% of the distance measured by tape measure between the two sites assessed. Time is the pulse wave travel time between common carotid and common femoral arteries.
Change in Baseline to Post-Treatment Indices of Cardiac Structure via Resting Echocardiography Imaging | Baseline; Post-treatment: 7 weeks after treatment initiation
  The ultrasound probe from the Terason 3000+ will then be used to capture standard parasternal short-axis, long-axis, apical and sub-sternal views of the heart. . Briefly, left ventricular mass and thickness, ejection fraction, left ventricular diastolic function, and left atrial volume index will be calculated.
Change in Baseline to Post-Treatment Central Augmentation Index | Baseline; Post-treatment: 7 weeks after treatment initiation
  The difference between early and late pressure peaks divided by pulse pressure
Change in Baseline to Post-Treatment Central Systolic blood pressure | Baseline; Post-treatment: 7 weeks after treatment initiation
  Blood pressure at the aorta close to the heart
Change in Baseline to Post-Treatment Central Pulse Pressure | Baseline; Post-treatment: one week after treatment completion; Follow-up for experimental group only: 8 weeks after post-treatment visit
  Change in the differences between central systolic and central diastolic pressures

CONTACTS AND LOCATIONS:
Overall Officials: Megan E Petrov, PhD, Principal Investigator — Arizona State University
Locations (1):
- Arizona State University, Phoenix, Arizona, United States